CLINICAL TRIAL: NCT01811680
Title: A Phase 1 Study of "An Exploratory Feasibility Clinical Study on a Variable Speed and Sensing Treadmill System (VASST) for Hemiparetic Gait Rehabilitation in Subacute Stroke Patients."
Brief Title: An Exploratory Clinical Study on a Variable Speed and Sensing Treadmill System (VASST) for Hemiparetic Gait Rehabilitation
Acronym: VASST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Chua Sui Geok, Karen, Principal Investigator, Tan Tock Seng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHG DSRB_D_2012/00571
Record Dates: First submitted 2013-03-05; First posted 2013-03-14 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Stroke; Hemiplegic Gait
Keywords: Stroke; Hemiplegia; Variable automated treadmill treadmill
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- supervised treadmill training (Experimental): Supervised treadmill training on variable sensing treadmill.
  Interventions: Device: Variable Speed and Sensing Treadmill

INTERVENTIONS:
Device: Variable Speed and Sensing Treadmill — open label study on variable speed and sending treadmill training for hemiplegic gait training.
  Other Names: VASST

SUMMARY:
To conduct a feasibility clinical trial to test a novel patient sensing automated treadmill device devised by local engineers for subacute hemiplegic stroke patients for gait rehabilitation. This is a phase 1 feasibility and safety trial on the above device for 10 chronic stroke patients with hemiparetic gait dysfunction to be conducted over a period of 2 months.

Research protocol and standardized outcomes measures will be used.

DETAILED DESCRIPTION:
To conduct a feasibility clinical trial to test a novel patient sensing automated treadmill device devised by local engineers for subacute hemiplegic stroke patients for gait rehabilitation. This device incorporates patient automated variable speeds and feedback, increased safety features with patient support harness and visual feedback providing ambulatory gait monitoring data. Methodology: 10 stable subacute hemiparetic stroke subjects will undergo supervised treadmill training using this device targeted at improving gait speed and walking independence. Outcomes will be measured at 4 time points pre and post training using clinical scales and temporal-spatial gait measurements. Importance of research to medicine: This study tests the possibility of patient initiated control and closed loop sensing feedback system to provide increased intensity, reduced risk of gait destabilisation and fall risk which are associated with current fixed treadmill training. Potential benefits with new device: Ability to train at self selected variable speeds including fast speeds, improved hemiplegic leg swing initiation and stride length, less assistance required from physiotherapist and reduced fall risk due to overhead safety harness and treadmill sensing and increased patient confidence. Possibility of ambulatory gait speed and force loading during treadmill training. Potential risks: Minor risks of fall are minimised as there is a safety harness and supervision by physiotherapist. Anticipated risks related to repetitive treadmill training with regards to cardiovascular and musculoskeletal side effects will be mitigated with strict patient inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. First ever stroke (ischaemic or haemorrhagic) confirmed on Computed Tomography or Magnetic Resonance imaging
2. Aged 21 - 80 years
3. Stroke duration of >3 months in outpatient phase (subacute -chronic stroke)
4. Able to walk overground at a self-selected speed of >0.2m/s with or without walking aids or lower limb orthoses for at least 150 meters with contact guard or supervision.
5. Functional ambulation category (FAC >/= 2) (Holden et al 1994)

Exclusion Criteria:

1. Cardiovascular conditions such as uncontrolled hypertension/hypotension, angina pectoris, recent myocardial infarction, congestive cardiac failure, known echocardiographic ejection fraction < 40% within 3 months of stroke, chronic arrhythmias (e.g. atrial fibrillation) within 3 months of study screening, pacemaker, uncontrolled Diabetes Mellitus.
2. End stage illness (advanced malignancy), pregnancy or end stage renal failure with life expectancy of <6 months.
3. Aphasia (inability to obey 2 step commands), communication disorder precluding understanding of instructions, cognitive impairment, dementia, untreated depression or psychiatric disorder.
4. Active lower limb arthritis, Pain (Visual Analogue Scale) >5/10, fixed orthopaedic deformities of the lower limb which would compromise safe ambulation on treadmill.
5. Moderate to severe lower limb spasticity or spasms (Modified Ashworth Scale >2)
6. Active trunk skin conditions, known abdominal aortic aneurysm, anticoagulation with warfarin precluding safe fit of gait harness

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chua Karen, MD, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- TTSH Rehab Medicine, Centre of Advanced Rehablitation Therapeutics (CART) , 11 Jalan Tan Tock Seng Hospital, Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supervised Treadmill Training
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Supervised Treadmill Training
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (9.85)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Singapore | 10

OUTCOME MEASURES:

1. Primary Outcome: 6 Minute Walk Test (Metres)
Description: 6 minute walk test - assess distance walked within 6 minutes as a sub maximal test of endurance (Assessed at weeks 0,2,4 and 8)
Time Frame: 8 weeks
Population: chronic stroke
Measure: Mean (Standard Deviation); unit: metres
Arm/Group | Supervised Treadmill Training
Number analyzed (Participants) | 10
metres | 54.3 (30.9)

2. Primary Outcome: 10 Meter Walk Test
Description: Assess time taken to walk 10meters to estimate walking speed(m/s) (Assessed at weeks 0,2,4,8)
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Supervised Treadmill Training
Number analyzed (Participants) | 10
m/s | 0.06 (0.07)

ADVERSE EVENTS:
Time Frame: 2 months
Groups:
- Supervised Treadmill Training: Research Intervention: Supervised treadmill training on variable sensing treadmill.
Arm/Group | Supervised Treadmill Training
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
There were technical limitations due to Gaitrite walkway malfunction midway in the trial leading to unreliable cadence results. Step length results were not affected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No